CLINICAL TRIAL: NCT06238687
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability , Pharmacokinetics and Preliminary Efficacy of STRO-002 in Chinese Adults With Advanced Epithelial Ovarian Cancer, Endometrial Cancer, and Other Advanced Malignant Solid Tumors.
Brief Title: A Study of STRO-002 in Chinese Adults With Epithelial Ovarian Cancer and Other Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Collaborators: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSL-B2276-1-01
Record Dates: First submitted 2023-11-21; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Neoplasm Malignant
Keywords: advanced malignant solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1(Phase I) (Experimental): STRO-002 3.5 mg/kg Open Lable
  Interventions: Biological: STRO-002
- Cohort 2(Phase I) (Experimental): STRO-002 4.3 mg/kg Open Lable
  Interventions: Biological: STRO-002
- Cohort 3(Phase I) (Experimental): STRO-002 5.2 mg/kg Open Lable
  Interventions: Biological: STRO-002
- Cohort A(Phase IIa) (Experimental): Recurrent and/or progressive ovarian epithelial cancer, confirmed by immunohistochemistry [IHC] testing with FolRα positive expression (TPS ≥ 75%).
  Interventions: Biological: STRO-002
- Cohort B(Phase IIa) (Experimental): Recurrent and/or progressive ovarian epithelial cancer, confirmed by IHC testing with FolRα positive expression (25% ≤ TPS < 75%).
  Interventions: Biological: STRO-002
- Cohort C(Phase IIa) (Experimental): Recurrent and/or progressive endometrial cancer, confirmed by IHC testing with FolRα positive expression (TPS ≥ 25%).
  Interventions: Biological: STRO-002
- Cohort D(Phase IIa) (Experimental): Recurrent and/or progressive non-small-cell lung cancer, confirmed by IHC testing with FolRα positive expression (TPS ≥ 25%).
  Interventions: Biological: STRO-002
- Cohort E(Phase IIa) (Experimental): Recurrent and/or progressive triple-negative breast cancer, confirmed by IHC testing with FolRα positive expression (TPS ≥ 25%).
  Interventions: Biological: STRO-002

INTERVENTIONS:
Biological: STRO-002 — STRO-002 is an Antibody-drug conjugates (ADCs) combine the specificity of monoclonal antibodies with the anti-tumor activity of cytotoxic drugs.

SUMMARY:
This is a multi-center, open-label, monotherapy dose escalation, PK bridging, and dose expansion Phase I/IIa study in Chinese adult subjects to evaluate the safety, tolerability, Pharmacokinetics (PK) profiles, immunogenicity, and preliminary efficacy of STRO-002 in patients with advanced malignant solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts, Phase I (dose escalation and PK bridging) and Phase IIa (dose expansion). Subjects in each cohort of Phase I will be administered 3 scheduled dose levels of STRO-002 as monotherapy by intravenous infusion until intolerable toxicity, radiographic disease progression, or subject withdrawal for other reasons. 5 dose arms are tentatively set based on the available safety, PK and efficacy data of STRO-002 for the Phase IIa (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy >3 months.
2. Subjects must have at least one measurable lesion (non-radiotherapy field) per RECIST v1.1.
3. The adverse reactions (ARs) of previous anti-tumor therapy must recover to NCI CTCAE v5.0 grade ≤ 1 (except for toxicity with no safety risks judged by investigators, such as alopecia).
4. For adequate bone marrow reserve and organ function.
5. Calculated QT interval corrected for heart rate using Fridericia correction formula (QTcF), screening and C1D1 predose ECG must be < 500 msec.
6. (Dose escalation + PK bridging)Relapsed and/or progressed at least one prior line of standard of care, or have no available standard of care, or are intolerable to standard of care, or have no further approved treatment options available.
7. (Dose expansion)For each cohort, the following criteria should be met: a. Cohorts A and B (ovarian cancer): High-grade serous epithelial ovarian cancer with a confirmed pathological diagnosis, fallopian tube cancer, or primary peritoneal carcinoma.b. Cohort C (endometrial cancer): Endometrial epithelial cancer with a confirmed pathological diagnosis (endometrioid adenocarcinoma; serous adenocarcinoma; undifferentiated carcinoma; mixed epithelial carcinoma; or adenocarcinoma not otherwise specified [N.O.S]), and the disease has relapsed or progressed after at least 1-line of platinum-based chemotherapy regimen or 1-line of immunotherapy-containing regimen, and no more than 3 lines of treatment regimen received previously. c. Cohort D (non-small-cell lung cancer): Unresectable locally advanced or metastatic non-small-cell lung cancer with a confirmed pathological diagnosis, and previous treatment meets the following criteria: - Patients without genetic mutations: If they receive 1-line platinumdoublet chemotherapy and anti-PD-1/PD-L1 combination at the same time, they have previously received at least 1-line treatment in the past and totally no more than 4 lines of treatment regimen; if they have received platinum-doublet chemotherapy sequentially and anti-PD-1/PD-L1, they have previously received at least 2-line treatment and totally no more than 4 lines of treatment regimen. - People with genetic mutations: Received at least 1-line approved targeted therapy, and previously no more than 4 lines of treatment regimen. d. Cohort E (triple-negative breast cancer): Unresectable locally advanced or metastatic breast cancer with a confirmed pathological diagnosis, and the ER, PR, and HER-2 are all negative. ER and PR negative are defined as: IHC ER < 1%, IHC PR < 1%. HER-2 negative is defined as: IHC HER-2 (-) or (1+). Patients with HER-2 (2+) must undergo FISH testing and the result is negative; they have previously received at least 1 line but no more than 4 lines of systemic anticancer therapy.

Exclusion Criteria:

1. Prior treatment with ADCs containing tubulin inhibitors (e.g., mirvetuximab of Immunogen, XMT-1536 of Mersana, which contains auristain derivatives that inhibit tubulin polymerization).
2. Previous treatment with other FolRα-targeting drugs.
3. History of severe allergy or anaphylactic reaction to monoclonal antibody therapy or antibody-related fusion protein treatment.
4. Prior anticancer therapy (prior to initial dose of study drug): Chemotherapy within 3 weeks, PARPi within 2 weeks, other therapeutic anticancer antibodies within 3 weeks, radio- or toxin-immunoconjugate (such as ADCs) within 10 weeks, Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 1 week, radion therapy/major surgery within 4 weeks (the definition of surgery refers to Grade 3-4 surgeries specified in the Measures for the Grade Management of Surgery in Medical Institutions issued by the National Health Commission of the PRC on December 06, 2022) or are in the recovery period from surgery (the investigator judges that there are still risks in participating the clinical study). 5. Pre-existing clinically significant ocular disorders including, but not limited to: Active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema and/or visual acuity reduced, Prior anticancer therapy (prior to initial dose of study drug): Chemotherapy within 3 weeks, PARPi within 2 weeks, other therapeutic anticancer antibodies within 3 weeks, radio- or toxin-immunoconjugate (such as ADCs) within 10 weeks, Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 1 week, radion therapy/major surgery within 4 weeks (the definition of surgery refers to Grade 3-4 surgeries specified in the Measures for the Grade Management of Surgery in Medical Institutions issued by the National Health Commission of the PRC on December 06, 2022) or are in the recovery period from surgery (the investigator judges that there are still risks in participating the clinical study).
5. Pre-existing clinically significant ocular disorders including, but not limited to: Active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema and/or visual acuity reduced, blurred vision, conjunctivitis, keratitis, cataracts with significant visual impairment, uveitis, Sjogren syndrome, and dry eye.

Patients who are required to take folic acid-containing supplements, e.g., folate deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT Assessment | From Day1 to Day21 after first dose of STRO-002
  Toxicity associated with the treatment of the investigational drug STRO-002.
AE Assessment | From first dose of STRO-002 until 28 days after the last dose of STRO-002
  The frequency of AE
AUC | From first dose of STRO-002 until 28 days after the last dose of STRO-002.
  PK parameter：area under the concentration-time curve (AUC)
Cmax | From first dose of STRO-002 until 28 days after the last dose of STRO-002.
  PK parameter：Cmax
Half life (t1/2) | From first dose of STRO-002 until 28 days after the last dose of STRO-002.
  PK parameter：half life (t1/2)
Overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1
Determine the recommended phase II dose (RP2D) | From first dose of STRO-002 until 28 days after the last dose of STRO-002.

SECONDARY OUTCOMES:
Occurrence of positive anti-drug antibodies (ADAs) and changes over time. | From first dose of STRO-002 until 28 days after the last dose of STRO-002.
  Occurrence of positive anti-drug antibodies (ADAs)
Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  DOR is defined as the time from the first documented response (CR or PR evaluated by RECIST v1.1) until the time of first documentation of disease progression by RECIST v1.1.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PFS is defined as a time from the first dose of STRO-002 to documented disease progression or death from any cause.
FolRα and cancer antigen 125 (CA-125) levels measured in tumor tissue | From first dose of STRO-002 until 28 days after the last dose of STRO-002.
  A CA-125 response is defined as at least a 50% reduction in CA-125 levels from a pretreatment sample, and the response must be confirmed and maintained for at least 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kongli zhu, Study Chair — Tasly Pharmaceutical Group Co., Ltd
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No